CLINICAL TRIAL: NCT01733914
Title: Phase II Study of Contralateral Acupuncture in the Treatment of Chronic Shoulder Pain
Brief Title: Contralateral Acupuncture in the Treatment of Chronic Shoulder Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Ming Yi, PhD, principle investigator, Dr, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007CB512501
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-05

CONDITIONS: Shoulder Pain
Keywords: shoulder pain; acupuncture
MeSH Terms: conditions — Shoulder Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Experimental group
  Interventions: Procedure: Acupuncture
- Waiting list (Sham Comparator): Control group
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture in the following acupoints on the contralateral side of pain site: Jiantong, Zhongzhu, Houxi, and Quchi. The patient will receive 5 treatments (each lasts 30 min) per week for four weeks.
  Arms: Acupuncture
Other: Control — Patients in the waiting list group received conventional orthopaedic therapy including physical exercise, heat or cold therapy. 50 mg diclofenac daily could be taken when the patient suffered from the pain. Injections or cortisone applications of any kind were not allowed.
  Arms: Waiting list

SUMMARY:
According to traditional Chinese medical theories, a variety of acupuncture formulas can treat diseases such as pain. For example, stimulating acupoints either local or distal to the pain site has been proposed under some conditions. We hypothesize that stimulating acupoints contralateral to the pain site can successfully treat chronic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Uni-lateral shoulder pain for 6 weeks to 2 years
* VAS score ≤ 50
* 25-65 years of age
* Positive Neer's or Hawkins' signs
* Accept the informed consent

Exclusion Criteria:

* Shoulder pain of neurological origins
* Shoulder pain of neck origins
* Systematic arthritis
* Wrist problems
* Previous shoulder, arm, neck or chest fractures or surgeries
* Mental diseases
* Pregnancy
* Inability to work for more than 3 months before treatment
* Diabetes
* Coagulative dysfunction
* Corticosterone or physicotherapy experience on the affected shoulder in the last 6 months
* Failure to accept the informed consent

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | before and 2, 4, 8 and 16 weeks after treatment start
  Pain assessment

SECONDARY OUTCOMES:
The MOS item short from health survey (SF-36) | before and 8 and 16 weeks after treatment start
  Quality of life assessment
Constant-Murley score | before and 2, 4, 8 and 16 weeks after treatment start
  shoulder motion score
DASH score | before and 2, 4, 8 and 16 weeks after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yi, PhD, Principal Investigator — Peking University
Locations (1):
- Province Hospital of Integrative Chinese and Western Medicine, Sichuan, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhang H, Sun J, Wang C, Yu C, Wang W, Zhang M, Lao L, Yi M, Wan Y. Randomised controlled trial of contralateral manual acupuncture for the relief of chronic shoulder pain. Acupunct Med. 2016 Jun;34(3):164-70. doi: 10.1136/acupmed-2015-010947. Epub 2016 Jan 21. PMID 26795764